CLINICAL TRIAL: NCT02197481
Title: BiClamp Forceps Liver Transection Versus Clamp Crushing Technique in Liver Resections: A Randomized Clinical Trial
Brief Title: Usefulness of BiClamp Forceps for Liver Resection: A Randomized Clinical Trial
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: The Second Hospital of Anhui Medical University (Other)
Collaborators: The First Affiliated Hospital of Anhui Medical University (Other)
Responsible Party: Principal Investigator, xpgeng, vice-president, The Second Hospital of Anhui Medical University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ahykdxdefsyy10
Record Dates: First submitted 2014-07-15; First posted 2014-07-22 (Estimated); Results first posted 2017-12-14 (Actual); Last update posted 2017-12-14 (Actual); Status verified 2017-05

CONDITIONS: Hepatobiliary Disease
Keywords: BiClamp forceps hepatectomy; Clamp crushing technique; Liver parenchyma transection; Randomized controlled trial
MeSH Terms: conditions — Digestive System Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Clamp-Crushing technique (Active Comparator): liver transection during hepatectomy by the routine clamp-crushing technical without BiClamp forceps assisted
  Interventions: Procedure: Clamp-Crushing technique
- BiClamp forceps hepatectomy (Experimental): The BiClamp forceps, a reusable bipolar sealing instrument for use in open surgery, was uniformly employed in all patients randomized to BiClamp forcep hepatectomy group in the present study.
  Interventions: Device: BiClamp forceps

INTERVENTIONS:
Procedure: Clamp-Crushing technique — Liver transection during hepatectomy by monopole electronicknife and blood vessel forceps, but without BiClamp forceps
  Arms: Clamp-Crushing technique
Device: BiClamp forceps — liver transection during hepatectomy by BiClamp forceps
  Arms: BiClamp forceps hepatectomy

SUMMARY:
The purpose of this study is to compare short-term and long-term efficacy of BiClamp forceps hepatectomy and clamp-crushing technique for parenchymal transection during elective hepatic resection.

DETAILED DESCRIPTION:
Background: Blood loss and the need for blood transfusions during the liver transection have shown to be correlated with higher morbidity and mortality rates and with worsen prognosis. Various devices of liver parenchymal transection have been developed with a view to reducing the intraoperative blood loss. However, to the present there is no randomized controlled trial evaluating the technique of BiClamp forceps during the liver transection. The goal of the present study was to evaluate the safety and effectiveness of BiClamp forceps transection in comparison to the clamp crushing technique in patients offered liver resection.

Intervention: One hundred patients with hepatobiliary disease need undergo hepatectomy at Anhui medical university were selected and divided into BiClamp forceps hepatectomy group and clamp-crushing hepatectomy group, each group contains 50 cases.

Results:

1. Clinical data include: blood loss during liver transection, total blood loss, blood transfusion, hospital stay, morbidity, mortality, biliary leakage, postoperative liver function, liver transection time, operation time, resection margins, need for portal trial clamping.
2. Statistical method: groups t-test, univariate/multivariate analysis, logistic regression analysis, mixed linear regression and Cox survival analysis were used.

ELIGIBILITY:
Inclusion Criteria:

* Both male and female, aged 18 or older
* Patients scheduled to undergo hepatic resection for some benign or malignant hepatobiliary disease
* Child-Pugh class A or B liver function
* BiClamp forceps hepatectomy and clamp-crushing feasible based on preoperative imaging
* No tumor invasion the main vein, hepatic artery and vein and major inferior vena cava
* No extrahepatic metastasis
* Voluntary participation in the study, and informed consent.

Exclusion Criteria:

* Age <18 years or> 65 years , pregnant or lactating women
* Preoperative liver function evaluation: Child-Pugh C grade
* Laparoscopic hepatectomy
* Extrahepatic metastasis
* Tumor invasion the main vein, hepatic artery and vein and major inferior vena cava
* The patient refused to sign the informed consent form

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 105 (Actual)
Dates: Start 2014-09; Primary Completion 2016-05 (Actual); Study Completion 2016-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Geng Xiaoping, Principal Investigator — The Second Hospital of Anhui Medical University
Locations (1):
- the Second Affiliated Hospital of Anhui Medical University, Hefei, Anhui, China

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Result] Kooby DA, Stockman J, Ben-Porat L, Gonen M, Jarnagin WR, Dematteo RP, Tuorto S, Wuest D, Blumgart LH, Fong Y. Influence of transfusions on perioperative and long-term outcome in patients following hepatic resection for colorectal metastases. Ann Surg. 2003 Jun;237(6):860-9; discussion 869-70. doi: 10.1097/01.SLA.0000072371.95588.DA. PMID 12796583
- [Result] Gurusamy KS, Pamecha V, Sharma D, Davidson BR. Techniques for liver parenchymal transection in liver resection. Cochrane Database Syst Rev. 2009 Jan 21;2009(1):CD006880. doi: 10.1002/14651858.CD006880.pub2. PMID 19160307
- [Result] Itoh S, Fukuzawa K, Shitomi Y, Okamoto M, Kinoshita T, Taketomi A, Shirabe K, Wakasugi K, Maehara Y. Impact of the VIO system in hepatic resection for patients with hepatocellular carcinoma. Surg Today. 2012 Dec;42(12):1176-82. doi: 10.1007/s00595-012-0306-6. Epub 2012 Sep 20. PMID 22993104
- [Derived] Chen JM, Geng W, Liu FB, Zhao HC, Xie SX, Hou H, Zhao YJ, Wang GB, Geng XP. BiClamp(R) forcep liver transection versus clamp crushing technique for liver resection: study protocol for a randomized controlled trial. Trials. 2015 Apr 30;16:201. doi: 10.1186/s13063-015-0722-1. PMID 25925431
- Available data/document: Study Protocol: PMID:25925431 — http://www.ncbi.nlm.nih.gov/pubmed/25925431

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Eligibility criteria included scheduled liver resection for benign or malignant hepatobiliary disease and a minimum age of 18 years.
Pre-assignment Details: Patients undergoing concomitant vascular resection or bile duct resection and those undergoing emergency liver resection were excluded.
Groups:
- Clamp-Crushing Technique: liver transection during hepatectomy by the routine clamp-crushing technical without BiClamp forceps assisted
  Clamp-Crushing technique: Liver transection during hepatectomy by monopole electric knife and blood vessel forceps, but without BiClamp forceps
Period: Overall Study
Arm/Group | Clamp-Crushing Technique | BiClamp Forceps Hepatectomy
Started | 43 (October 2014) | 43
Completed | 43 (February 2016) | 43
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Clamp-Crushing Technique | BiClamp Forceps Hepatectomy | Total
Number analyzed (Participants) | 43 | 43 | 86
Age, Continuous [Mean (Standard Deviation); unit: years] | 53.12 (10.84) | 55.98 (11.30) | 54.55 (11.10)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 16 | 23 | 39
  Male | 27 | 20 | 47
Region of Enrollment [Number; unit: participants]
  China | 43 | 43 | 86
Transection surface area [Mean (Standard Deviation); unit: cm2] | 69.11 (40.09) | 65.16 (44.30) | 67.14 (42.04)
Specimen weight [Mean (Standard Deviation); unit: g] | 230.73 (191.35) | 193.25 (182.48) | 211.99 (186.82)

OUTCOME MEASURES:

1. Primary Outcome: The Total Blood Loss
Description: Blood loss during operation. Blood loss was calculated from the beginning to the end of operation The amount of blood loss was measured from the suction volume after subtraction of rinse fluids and from the weight of soaked gauzes that were used during transection
Time Frame: an expected average of 80 minutes
Measure: Mean (Standard Deviation); unit: ml
Arm/Group | Clamp-Crushing Technique | BiClamp Forceps Hepatectomy
Number analyzed (Participants) | 43 | 43
ml | 376.73 (303.67) | 339.81 (257.20)

2. Secondary Outcome: Liver Transection Time
Description: liver transection time was calculated from the beginning to the end of the liver resection
Time Frame: an expected average of 40 minutes
Measure: Mean (Standard Deviation); unit: min
Arm/Group | Clamp-Crushing Technique | BiClamp Forceps Hepatectomy
Number analyzed (Participants) | 43 | 43
min | 25.51 (12.19) | 26.21 (17.17)

3. Secondary Outcome: Mortality
Description: Operative mortality was defined as any death resulting from a complication during surgery
Time Frame: 90 days
Measure: Number; unit: participants
Arm/Group | Clamp-Crushing Technique | BiClamp Forceps Hepatectomy
Number analyzed (Participants) | 43 | 43
participants | 0 | 0

4. Secondary Outcome: Morbidity
Time Frame: 90 days
Measure: Number; unit: participants
Arm/Group | Clamp-Crushing Technique | BiClamp Forceps Hepatectomy
Number analyzed (Participants) | 43 | 43
participants | 13 | 12

5. Secondary Outcome: Biliary Leakage
Description: Biliary leakage was documented in line with the International Study Group of Liver Surgery (ISGLS) definitions and grading systems
Time Frame: 90 days
Measure: Number; unit: participants
Arm/Group | Clamp-Crushing Technique | BiClamp Forceps Hepatectomy
Number analyzed (Participants) | 43 | 43
participants | 4 | 2

6. Secondary Outcome: Duration of Postoperative Hospital Stay
Description: Time from day of operation to day of discharge
Time Frame: an expected average of 12 days
Measure: Mean (Standard Deviation); unit: days
Arm/Group | Clamp-Crushing Technique | BiClamp Forceps Hepatectomy
Number analyzed (Participants) | 43 | 43
days | 8.65 (2.02) | 8.81 (2.49)

7. Secondary Outcome: Number of Participants Requiring a Blood Transfusion
Description: Administration of blood transfusions is documented for the intraoperative and postoperative period until 48 hours postoperatively
Time Frame: 2 days
Measure: Number; unit: participants
Arm/Group | Clamp-Crushing Technique | BiClamp Forceps Hepatectomy
Number analyzed (Participants) | 43 | 43
participants | 2 | 4

8. Secondary Outcome: Total Bilirubin
Description: serum total bilirubin on 3 postoperative day (umol/L)
Time Frame: 3 postoperative day
Measure: Mean (Standard Deviation); unit: umol/l
Arm/Group | Clamp-Crushing Technique | BiClamp Forceps Hepatectomy
Number analyzed (Participants) | 43 | 43
umol/l | 17.70 (11.34) | 18.46 (17.75)

ADVERSE EVENTS:
Arm/Group | Clamp-Crushing Technique | BiClamp Forceps Hepatectomy
Serious Adverse Events (participants affected / at risk) | 4/43 | 2/43
Other Adverse Events (participants affected / at risk) | 12/43 | 12/43
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Clamp-Crushing Technique (N=43) | BiClamp Forceps Hepatectomy (N=43)
biliary leakage (Hepatobiliary disorders) | 3 (43) | 1 (43) — percutaneous drainage
pleural effusions (General disorders) | 1 (1) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 2% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Clamp-Crushing Technique (N=43) | BiClamp Forceps Hepatectomy (N=43)
pleural effusions (General disorders) | 7 (7) | 7 (7)
Liver failure (Hepatobiliary disorders) | 2 (2) | 2 (2)
Wound infection (Infections and infestations) | 2 (2) | 2 (2)
Biliary leakage (Hepatobiliary disorders) | 1 (1) | 1 (1)

LIMITATIONS AND CAVEATS:
Owing to the small number of patients, no subgroup analysis based in type of hepatic resection or hepatic portal occlusion, So it is unclear whether the advantage of BiClamp® forceps is applicable to special type hepatic resection subgroups.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes